CLINICAL TRIAL: NCT02364830
Title: Randomised Clinical Trial: Enteric-coated Anise-oil Capsules vs. Placebo & Active Controlled in Irritable Bowel Syndrome - A 4 Week Double-blind Study With 2 Weeks Follow-up
Brief Title: Clinical Effectiveness of Enteric Coated(E.C.) Anise-oil on Irritable Bowel Syndrome
Acronym: IBS-Anise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Maryam Mosaffa-Jahromi, PharmD., PhDc of Traditional Pharmacy, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E.C. Anise-oil on IBS; Dr.Mosaffa (Registry Identifier: Dr.Mosaffa)
Record Dates: First submitted 2015-02-05; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Pimpinella anisum L.; Peppermint oil; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anise-oil EC (Active Comparator): Intervention Group: Anise-oil EC Capsule,One Cap(187mg)/day for 4 weeks. Patients will be Followed at Baseline, 4 and 6 Weeks after Starting Intervention.
  Interventions: Drug: Anise-oil EC Capsule
- Placebo (Placebo Comparator): Placebo Group: One Placebo Capsule/Day for 4 Weeks. Patients Will be Followed at Baseline, 4 and 6 Weeks after Starting Intervention.
  Interventions: Other: Placebo
- Colpermin® (Active Comparator): Colpermin® Group: One Colpermin® Capsule/Day for 4 Weeks. Patients Will be Followed at Baseline, 4 and 6 Weeks after Starting Intervention.
  Interventions: Drug: Colpermin®

INTERVENTIONS:
Drug: Anise-oil EC Capsule — Anise-oil EC Capsule,One Cap(187mg)/day for 4 Weeks
  Other Names: Group A
  Arms: Anise-oil EC
Other: Placebo — One Placebo Capsule/Day for 4 Weeks
  Other Names: Group B
  Arms: Placebo
Drug: Colpermin® — Colpermin® Capsule/Day for 4 Weeks
  Other Names: Group C
  Arms: Colpermin®

SUMMARY:
Colpermin ® (Peppermint oil) is used in the treatment of Irritable Bowel Syndrome but Peppermint (Mentha x piperita) isn't native in Iran. So in this study the Enteric-Coated of Anise-oil will formulate and use in treatment of Irritable Bowel Syndrome with pain and bloating.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of Enteric-coated Anise-oil capsules comparing with placebo and Colpermin® for treatment of IBS patients. 120 patients with confirmed IBS with non-response criteria selected. In this double blind pilot study, the patients and researchers will be blinded about Receiving Drug, Placebo and Active allocation. Patients will be randomized into group A (Anise-oil EC Capsule 187 mg daily, for 4 weeks), group B (placebo Capsule once daily, for 4 weeks) and group B (Colpermin® Capsule once daily, for 4 weeks). At the end of therapy (4 weeks) and at baseline (first), 2 weeks after receiving drug, placebo and Colpermin® IBS load, will be evaluated and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the Rome III Modular Questionnaire
* Patients with 50 years were required to have a colonoscopy performed within the previous 5 years
* Patients under the age of 50 years were required to have a sigmoidoscopy performed

Exclusion Criteria:

* Unable or unwilling patients to use an acceptable method of birth control
* Pregnant or nursing females
* Previous gastrointestinal or abdominal surgery (except for common causes unrelated to IBS)
* Organic disorder of the large or small bowel (e.g. ulcerative colitis, Crohn's disease)
* Mechanical obstruction
* Unexplained significant weight loss or rectal bleeding
* Diagnosis of any medical condition associated with constipation (other than IBS)
* Cancer
* Abnormal laboratory tests
* Abuse of alcohol or drugs

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Composite of Quality of Life (QOL), pain, flatulence, diarrhea, constipation, reflux, headache and tiredness | Baseline
  (IBS-QOL) questionnaire and 10-point visual scale ranging

SECONDARY OUTCOMES:
Composite of Change in Quality of Life (QOL), pain, flatulence, diarrhea, constipation, reflux, headache and tiredness at end of treatment | 4 weeks after start treatment
  (IBS-QOL) questionnaire and 10-point visual scale ranging
Composite of Change in Quality of Life (QOL), pain, flatulence, diarrhea, constipation, reflux, headache and tiredness at end of treatment | End of Follow Up(6 weeks after staring intervention)
  (IBS-QOL) questionnaire and 10-point visual scale ranging

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Mosaffa-Jahromi, PhDc, Principal Investigator — Department of Traditional Pharmacy, School of Pharmacy and Pharmaceutical Sciences Research Center, Shiraz University of Medical Sciences, Shiraz, Iran
Locations (2):
- Iran (2):
  - Dr. Kamran Bagheri Lankarani, Shiraz, Fars
  - Dr. Maryam Mosaffa-Jahromi, Shiraz, Fars